CLINICAL TRIAL: NCT00634192
Title: A Multicenter, Open Label, 2 Period Cross-over Study to Evaluate the PK of a 8 Week Continuous Treatment With 1x300mg/d and 2x300mg/d Tobramycin Inhaled With a 'Soft Mist' Nebulizer in Cystic Fibrosis (CF) Subjects
Brief Title: Pharmacokinetic Evaluation of an 8 -Week Treatment With Inhaled Tobramycin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CTBM100DDE01
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Pseudomonas Infections
Keywords: Chronic infection with P. aeruginosa in Cystic Fibrosis subjects
MeSH Terms: conditions — Pseudomonas Infections | interventions — Tobramycin

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: tobramycin
- 2 (Experimental)
  Interventions: Drug: tobramycin

INTERVENTIONS:
Drug: tobramycin — 1x300mg/d inhaled
  Arms: 1
Drug: tobramycin — 2x300mg/d inhaled
  Arms: 2

SUMMARY:
This study is designed to provide data about the pharmacokinetics (PK), safety and tolerability of two continuous treatment regimes of tobramycin nebulized solution delivered via a 'soft mist' nebulizer in Cystic Fibrosis (CF) subjects. Each treatment period will last 8 weeks. Additionally the PK of patients with a normal forced expiratory flow in 1 second (FEV1) (FEV1≥80% predicted) will be compared to patients with an abnormal FEV1 (FEV1<80% predicted).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged ≥6 years at the time of screening, with an Informed Consent Form signed by patient and if appropriate by parent/legal guardians, prior to any study-related procedure.
* Confirmed diagnosis of CF by the presence of one or more clinical features of CF in addition to a quantitative pilocarpine iontophoresis sweat chloride test of >60 mEq/L; or identification of well-characterized disease-causing mutations in each CFTR gene; or an abnormal nasal transepithelial potential difference characteristic of CF.
* P aeruginosa must be present in sputum or deep throat swab (or bronchoalveolar lavage [BAL]) at the screening visit and within 6 months prior to screening.

Exclusion Criteria:

* History of sputum (or BAL) culture yielding Burkholderia cepacia (B cepacia) within 2 years prior to screening and/or sputum culture yielding B cepacia at screening.
* FEV1 <25% of normal predicted values for age, sex, and height based on Knudson criteria at screening.
* Hemoptysis of more than 60 cc at any time within 30 days prior to study drug administration.
* Known local or systemic hypersensitivity to aminoglycosides or inhaled antibiotics.
* GFR<60ml/min/1.73m2 calculated with the Formula by Schwartz, BUN 40 mg/dl or more, or an abnormal urinalysis defined as 2+ or greater proteinuria.
* History of tinnitus or pathologic audiometry
* diagnosis of Allergic bronchopulmonary aspergillosis (ABPA) at screening
* Initiation of treatment with macrolide antibiotics within 28 days prior to study drug administration (subjects may be taking macrolide antibiotics at the time of enrollment, but they must have initiated treatment at least 28 days prior to study drug administration).
* Use of loop diuretics within 7 days prior to study drug administration.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 6 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-02 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the serum pharmacokinetics (PK) of inhaled tobramycin (AUC 0-90') of continuous daily dosing regimens with 2x300mg/d Tobramycin Nebuliser Solution (=TNS) inhaled with the PARI eFlow® rapid in Cystic Fibrosis (CF) subjects | 8 wks

SECONDARY OUTCOMES:
Serum PK of inhaled tobramycin (AUC 0-90') of continuous daily dosing regimens with 1 x 300mg/d tobramycin nebulized solution (= TNS) inhaled with the PARI eFlow rapid in cystic fibrosis subjects. | 8 wks
Compare serum PK of inhaled tobramycin (trough-/peak-level)of both dosing regimens in CF-subjects with a FEV1≥80% vs. CF-Subjects with a FEV1<80%. | 8 weeks
Change of MIC of P. aeruginosa during a continuous treatment with 1 x 300 mg/d and 2 x 300 mg/d TNS. | 8 weeks
Assess safety of a continuous daily dosing regimen with 1 x 300 mg/d and 2 x 300 mg/d TNS over 8 weeks, compared to historic safety data of the 4 week on/off dosing regimen with 2 x 300 mg/d. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma AG, Study Chair — Novartis Pharmaceuticals
Locations (8):
- Germany (8):
  - Novartis Investigator Site, Berlin
  - Novartis Investigator Site, Cologne
  - Novartis Investigator Site, Frankfurt
  - Novartis Investigator site, Halle
  - Novartis Investigator Site, Hamburg
  - Novartis Investigator Site, Hanover
  - Novartis Investigator Site, Heidelberg
  - Novartis Investigator Site, Munich

REFERENCES:
- [Result] van Koningsbruggen-Rietschel S, Heuer HE, Merkel N, Posselt HG, Staab D, Sieder C, Ziegler J, Krippner F, Rietschel E. Pharmacokinetics and safety of an 8 week continuous treatment with once-daily versus twice-daily inhalation of tobramycin in cystic fibrosis patients. J Antimicrob Chemother. 2016 Mar;71(3):711-7. doi: 10.1093/jac/dkv399. Epub 2015 Nov 30. PMID 26626719